CLINICAL TRIAL: NCT06780761
Title: Infant Simulator Training to Measure Pediatric Vital Signs
Acronym: PedVit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hatice Uzşen, Principal investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022-577
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Vital Signs; Simulation Training
Keywords: vital sign; pediatric; nursing; simulation

STUDY DESIGN:
Intervention Model Description: The author further demonstrated taking body temperature, heart rate and its characteristics, respiratory rate and saturation, blood pressure and pain assessment in line with previously created cases on the NOELLE® Maternal Birthing Simulator with Advanced Resuscitation Neonatal M-W45111 to the students deployed in the intervention group
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and biostatisticians were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Students were trained about taking body temperature, heart rate and its characteristics, respiratory rate and saturation, blood pressure, and pain assessment in line with previously created cases on the NOELLE® Maternal Birthing Simulator with Advanced Resuscitation Neonatal M-W45111.
  Interventions: Other: simulation training
- Control (Active Comparator): Students were trained on how to measure the five vital signs, which tools to use and why, and normal and abnormal vital sign values by demonstration and explanation on a pediatric nursing manikin.
  Interventions: Other: Classical training

INTERVENTIONS:
Other: simulation training — The author further demonstrated taking body temperature, heart rate and its characteristics, respiratory rate and saturation, blood pressure and pain assessment in line with previously created cases on the NOELLE® Maternal Birthing Simulator with Advanced Resuscitation Neonatal M-W45111 to the students deployed in the intervention group. Furthermore the students were allowed to work individually on the infant simulator, their questions were answered and feedback was given to them. Students were also offered free time to work on the infant simulator. One week after the training, before proceeding with the clinical practice, the students were individually assessed on measuring the vital signs by 2 different observers and were administered the post-tests.
  Arms: intervention
Other: Classical training — Before proceeding with the clinical practice, the students deployed in the control group were trained on how to measure the five vital signs, which tools to use and why, and normal and abnormal vital sign values by demonstration and explaining on a pediatric nursing manikin. Then, volunteering students were given the opportunity to develop their vital sign measurement skills on a pediatric nursing manikin and feedback was provided to them. One week after the training, all students were individually assessed on measuring the vital signs by 2 different independent observers on the simulator neonatal used in the intervention group and they were administered the post-tests.
  Arms: Control

SUMMARY:
Providing training to nursing students in the field of pediatric care requires having the competencies to care for the pediatric population. However, as the margin of error in pediatric care is quite narrow, nursing students need to undertake a comprehensive laboratory practice before implementing their care skills unsupervised in the pediatric ward. Nursing students can develop their professional skills by gaining the necessary confidence and skills with simulation methods.

DETAILED DESCRIPTION:
Simulation makes possible for students to feel a pulse, observe chest movements, hear respiration sounds, measure blood pressure, and evaluate results, thus allowing students to practice with concrete examples of various conditions. Hence simulation-based training, one of the important learning techniques, is assumed to help nursing students overcome the difficulties they will experience in measuring the children's vital signs

ELIGIBILITY:
Inclusion Criteria:

* Having taken the Pediatric Nursing course
* Voluntarily participating in the study

Criteria for exclusion from the study were as follows:

* Failure to complete the research process
* Filling out the necessary forms incompletely

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Vital Signs Scale (V-Scale) | It was assessed just before training as baseline. When all training was completed, ıt was assessed after 1 week again.
  The scale, originally developed by Mok et al. in 2015, was further adapted to Turkish by Ertuğ (2018). The 5-point Likert-type scale consists of 16 items and 5 factors. The sub-scales are workload, technology, communication, knowledge and key indicators. The total score varies between 16 and 80. A low score indicates that nurses have a low attitude towards vital signs monitoring while a higher score indicates a positive attitude towards vital signs monitoring. T

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Scale | When simulation based training was completed, ıt was assessed after 1 week.
  The scale originally published by the National Nursing Association was adapted to Turkish by Karaçay and Kara in 2017. The scale, widely used to measure students' attitudes and beliefs about simulation, consists of 13 items and 2 sub-scales

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Uzşen, Phd, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Black Sea Zone, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No